CLINICAL TRIAL: NCT00115206
Title: A Pilot Study of the Effects of Neutropenia on Patient Reported Outcomes During Chemotherapy With or Without Neulasta® (Pegfilgrastim) in Subjects With Advanced NSCLC
Brief Title: Neulasta® in Subjects With Advanced Non-Small-Cell Lung Cancer (NSCLC) During Chemotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20020121
Record Dates: First submitted 2005-06-21; First posted 2005-06-22 (Estimated); Last update posted 2009-04-06 (Estimated); Status verified 2009-04

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; NSCLC; Fever; Neutropenia; Neulasta®; Quality of Life; Chemotherapy; Amgen
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Fever; Neutropenia | interventions — pegfilgrastim

INTERVENTIONS:
Drug: Neulasta® (pegfilgrastim)

SUMMARY:
The purpose of this study is to estimate the relationship between patient reported outcomes (PROs) and neutropenia (or its complications) in NSCLC subjects receiving chemotherapy with or without Neulasta® (pegfilgrastim).

ELIGIBILITY:
Inclusion Criteria: - Non-small cell lung cancer, not previously treated with chemotherapy or radiotherapy - ECOG performance status 0 or 1 - ANC greater than or equal to 2.0 x 10^9/L Exclusion Criteria: - Cancer other than NSCLC within 5 years of enrollment, with the exception of surgically cured basal cell carcinoma or in situ carcinoma of the cervix - Treatment less than or equal to 30 days prior with any experimental agent - Subjects with symptomatic brain metastases - Subject is currently enrolled or has not yet completed at least 30 days since ending other investigational device or drug trial(s) or is receiving other investigational agent(s)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-07; Study Completion 2004-07

PRIMARY OUTCOMES:
Quality of Life

SECONDARY OUTCOMES:
Quality of Life, *Neutropenia, *Hospitalization, *Disease Response

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: FDA-approved Drug Labeling — http://www.neulasta.com/